CLINICAL TRIAL: NCT06471283
Title: Contribution of Physical Activity Per Dialytic in Chronic Dialysis Patients
Brief Title: Contribution of Per Dialytic Physical Activity in Chronic Dialysis Patients
Acronym: ACTIDIAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal André Grégoire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GHT_CHIM_RIRCM20220613
Record Dates: First submitted 2024-05-29; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-05

CONDITIONS: Dialysis
Keywords: dialysis patients; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group. This group will practice physical activity during dialysis sessions. (Experimental): Exercise using the LEMCO Hospital Bed Pedal Exerciser during dialysis.
  Interventions: Other: physical activity

INTERVENTIONS:
Other: physical activity — Exercising physical activity during dialysis
  Other Names: practice of physical activity during dialysis sessions

SUMMARY:
Dialysis patients have reduced walking capacity and an important risk of high blood pressure. These complications are associated with a decline in quality of life and increased mortality. The hypothesis of the study is to show that physical activity during the dialysis session in dialyzed patients has a benefit on quality of life, as well as on muscle, cardiovascular and dialysis parameters.

DETAILED DESCRIPTION:
Dialysis patients have reduced aerobic capacity, walking ability, and an increased risk of hypertension. These complications are associated with a decline in quality of life and increased mortality.

Since asthenia is too intense after the dialysis session, patients are encouraged to perform physical activity during dialysis sessions. Some studies have shown that physical activity during dialysis can have benefits on quality of life and improve muscle parameters, but without this being clinically significant. Other studies show no benefit. The objective of the study is to explore the benefits of physical activity on quality of life, muscle parameters, and biological and dialysis parameters in a cohort of compliant hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over, undergoing chronic hemodialysis at CHI André Grégoire for more than 3 months.
* Consent to participate in physical activity during dialysis sessions.
* Written informed consent.
* Affiliation with a social security system

Exclusion Criteria:

* Lower limb amputation without a prosthesis.
* Non-healed foot wounds.
* Hemoglobin < 8 g/dl.
* Patient refusal to participate.
* Severe respiratory (oxygen dependence) or cardiac disease (NYHA class 3 or 4, LVEF < 30%).
* Advanced dementia or psychiatric illness impeding cooperation, or refusal to consent.
* Non-French speaking patients unable to understand the study.
* Patients under guardianship.
* Advanced osteoarthritis, recent hip or knee prosthesis (< 3 months).
* Hypotension (BP < 90/40 mmHg) or hypertension (BP > 180/110 mmHg).
* Fever (temperature >= 38°C).
* Hypoglycemia (fingerstick glucose < 0.8 g/l) in diabetic patients.
* Dyspnea or desaturation in ambient air < 95%.
* COVID-19 symptoms within the last 21 days, positive PCR test, unable to pedal.
* Chest pain or unstable angina.
* Muscle or joint contraindications to the pedal exerciser as assessed by a physiotherapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in the quality of life of patients | 17 weeks
  Score of the Short Form-36 (SF36) questionnaire. The SF36 score varies from 0 to 100. A low score reflects a perception of poor health, loss of function, and presence of pain.
  A high score reflects a perception of good health, an absence of functional deficit and pain.

SECONDARY OUTCOMES:
Change in dialysis parameters (KT/V= clearance time/volume) | 17 weeks
  measurement of clearance time/volume (KT/V)
Change in muscle parameters | 17 weeks
  Score of the Medical research council scale (MRC)
Change in nutritional parameters | 17 weeks
  Measurement of body mass index (BMI)
Change in inflammatory parameters | 17 weeks
  measurement of CRP
Change in lipid profile | 17 weeks
  Measurement of total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides
Change in blood pressure | 17 weeks
  Measurement of systolic and diastolic blood pressure
Change in heart rate | 17 weeks
  measurement of pulse
Change in glycemic control | 17 weeks
  Levels of albumin
Change in glycemic control | 17 weeks
  Levels of prealbumin

CONTACTS AND LOCATIONS:
Overall Officials: Marion GAUTHIER, Principal Investigator — Centre Hospitalier Intercommunal André Grégoire
Locations (1):
- CHI Andre Gergoire, Montreuil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho JH, Lee JY, Lee S, Park H, Choi SW, Kim JC. Effect of intradialytic exercise on daily physical activity and sleep quality in maintenance hemodialysis patients. Int Urol Nephrol. 2018 Apr;50(4):745-754. doi: 10.1007/s11255-018-1796-y. Epub 2018 Jan 23. PMID 29362960
- [Background] Assimon MM, Wang L, Flythe JE. Intradialytic Hypertension Frequency and Short-Term Clinical Outcomes Among Individuals Receiving Maintenance Hemodialysis. Am J Hypertens. 2018 Feb 9;31(3):329-339. doi: 10.1093/ajh/hpx186. PMID 29077786